CLINICAL TRIAL: NCT03392233
Title: A Phase II Study to Evaluated the Long-term of Safety and Efficacy of Stereotactic Body Radiation Therapy for Spinal Metastases in Favorite Tumors
Brief Title: Stereotactic Body Radiation Therapy for Spinal Metastases in Favorite Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT-001
Record Dates: First submitted 2017-12-31; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer; Prostate Cancer; Non Small Cell Lung Cancer
Keywords: spinal metastases; Stereotactic body radiation therapy(SBRT); breast cancer; prostate cancer; non small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Eligible patients will receive Stereotactic body radiation therapy (SBRT) for spinal metastatic lesion in 24Gy/3f(cervical vertebra) or 30Gy/3f (thoracic vertebra/lumbar vertebra) every other day and receive relevant system treatment at same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase II open lable Study (Experimental): Eligible patients will receive Stereotactic body radiation therapy (SBRT) for spinal metastatic lesion in 24Gy/3f(cervical vertebra) or 30Gy/3f (thoracic vertebra/lumbar vertebra) every other day and receive relevant system treatment at same time.
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Eligible patients will receive Stereotactic body radiation therapy (SBRT) for spinal metastatic lesion in 24Gy/3f(cervical vertebra) or 30Gy/3f (thoracic vertebra/lumbar vertebra) every other day and receive relevant system treatment at same time

SUMMARY:
Stereotactic Body Radiation Therapy(SBRT) for spinal metastases has been proved a good results in pain relieve and local control, However,the longterm of efficacy and safety of this regimen is unclear.The purpose of the study is to evaluate the longterm outcome of this therapeutic regimen in selective patients who will be survival more than 2 years.

DETAILED DESCRIPTION:
Recently,Stereotactic Body Radiation Therapy(SBRT) become an alternative regimen for spinal metastases due to it's high dose cover the metastatic lesion and low dose in the adjacent spinal cord which result in more efficacy and less toxicity. However,the longterm of efficacy and safety of this regimen is unclear because of shortly median survival among unselective spinal metastases.To our knowledge,the median survival of some favorite metastatic diseases will be more than two years if they received appropriate system therapy.these include hormones dependent brest cancer/prostate cancer,and EGFR mutation non-small cell lung cancer(NSCLC) ect.The purpose of the study is to evaluate the longterm outcome of this therapeutic regimen in selective patients who will be survival more than 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. WHO scores 0-2;
2. The primary lesion was confirmed by pathology or cytology;
3. The metastatic lesions were diagnosed by imaging(CT,MRI,PET-CT,ECT),or the lesions were confirmed by biopsy;
4. The metastatic lesion was limited in 3 consecutive vertebral bodies;
5. The baseline pain score was ≥5(NRPS) and the use of analgesic drugs was recorded;
6. The enhanced MRI scan of involved vertebral bodies was required in the 2 weeks before radiotherapy;

Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

1. Leukocytes ≥ 3.0 x109/ L;
2. Absolute neutrophil count (ANC) ≥ 1.5 x109/ L;
3. Platelet count ≥ 100 x109/ L;
4. Hemoglobin (Hb) ≥ 9g/ dL;
5. Total bilirubin ≤1.5 x the upper limit of normal (ULN);
6. Alanine aminotransferase (ALT) ≤ 3 x ULN;
7. Aspartate aminotransferase (AST) ≤ 3 x ULN;
8. Serum creatinine ≤ 1.5 x the ULN;
9. Signed informed consent;

Exclusion Criteria:

1. There were significant changes in the shape of the vertebral body (the height of the vertebral body was compressed≥ 50%) or the vertebral body was unchanged but the volume of the dissolving bone was≥ 50% and could lead to serious bone adverse events;
2. There were >3 consecutive vertebral bodies involved;
3. Spinal cord compression has occurred;
4. The gap between tumor and spinal cord was less than 3mm;
5. The metastatic area previously received radiation;
6. Pregnant and Nursing women;
7. Uncontrolled co-morbid illnesses;

9.refused to signed informed consent;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-08-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of relieve pain | One week after radiation to 2 years late
  According to the Numerical Rating Pain Scale (NRPS)

SECONDARY OUTCOMES:
The degree of relieve pain | One week after radiation to 2 years late
  According to the Numerical Rating Pain Scale (NRPS)
The duration relieve pain | One week after radiation to 2 years late
  According to the Numerical Rating Pain Scale (NRPS)
The incidence of toxicity | One week after radiation to 2 years late
  Common Terminology Criteria for Adverse Events v3.0 (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Ming Ye, Master, Principal Investigator — Department of Radiation Oncology,Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine
Locations (1):
- Department of Radiation Oncology,Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China